CLINICAL TRIAL: NCT06219876
Title: Comparison of the Efficacy of High Intensity Laser Therapy and Low Level Laser Therapy in the Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Handan Elif Nur BAYRAKTAR, Dr., Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1254
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome; Electromyography; Low-Level Laser Therapy; Ultrasound Imaging
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): wrist splints of an appropriate size in a neutral position for at least 8 hours at night for 3 months
  Interventions: Other: wrist splint
- Low Level Laser Treatment (Active Comparator): * wrist splints of an appropriate size in a neutral position for at least 8 hours at night for 3 months
  * received an additional LLLT
  Interventions: Device: low level laser treatment
- High Intensity Laser Treatment (Active Comparator): * wrist splints of an appropriate size in a neutral position for at least 8 hours at night for 3 months
  * received an additional HILT
  Interventions: Device: High intensity laser treatment

INTERVENTIONS:
Device: low level laser treatment — The laser device from Mectronic Medicale was used for LLLT. LASER treatments were to be performed every other day for a total of 10 sessions.
  Arms: Low Level Laser Treatment
Device: High intensity laser treatment — The laser device from HIRO TT (ASA, Italy) was used for HILT. LASER treatments were to be performed every other day for a total of 10 sessions.
  Arms: High Intensity Laser Treatment
Other: wrist splint — wrist splints of an appropriate size in a neutral position for at least 8 hours at night for 3 months
  Arms: Control

SUMMARY:
Carpal tunnel syndrome is the most common entrapment neuropathy and is frequently encountered in clinical practice. Although there is no standard protocol for its treatment, conservative treatment methods are preferred. In our study, we aimed to clinically compare the efficacy of high and low intensity laser treatments in patients with carpal tunnel syndrome. By using methods such as electromyography and ultrasound, we aimed to provide a more objective evaluation

DETAILED DESCRIPTION:
Our study was designed as a prospective, randomised, controlled, single-centre trial. A total of 63 patients aged 18-65 years with electrophysiologically diagnosed mild to moderate carpal tunnel syndrome and 114 hands were included in the study. Patients were divided into 3 groups. Patients in all three groups wore a neutral wrist splint of appropriate size. The second group included patients who additionally received low level laser therapy (LLLT), and the third group included patients who additionally received high intensity laser therapy (HILT). All groups underwent clinical, electrophysiological, and ultrasonographic examinations at the beginning of the treatment, at 1st month, and at 3rd month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 65 years
2. Mild CTS (sensory conduction velocity at the second finger wrist < 41.26 m/sec, motor distal latency < 3.60 msec) or Moderate CTS (sensory conduction velocity at the second finger wrist < 41.26 m/sec and motor distal latency > 3.60 msec) according to the electrophysiological data were included in the study.

Exclusion Criteria:

1. Patients with local (osteophytes, ganglion cysts, lipomas, muscle and tendon abnormalities, etc.) and systemic (diabetes mellitus, acromegaly, hypothyroidism, pregnancy, etc.) diseases causing symptoms were included in the study.) causing CTS,
2. Patients who underwent surgical treatment for CTS
3. Patients who received injections for CTS in the last 6 months
4. Patients diagnosed with severe CTS on EMG (SAP not obtained in sensory conduction studies and/or CMAP < 5 mV in motor conduction studies)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
The Boston Symptom Severity Scale (BSSS) | end of 1. month
  The Boston Symptom Severity Scale consists of 11 questions, with each question scored between 1 and 5. The average score is calculated by summing the points received for each problem and dividing by the number of questions. A high score indicates that symptoms are severe and functional capacity is limited. The maximum score on this scale is 55 and the minimum score is 11.
The Boston Functional Capacity Scale (BFCS) | end of 1. month
  The Boston Functional Capacity Scale consists of 8 questions, with each question scored between 1 and 5. The average score is calculated by summing the points received for each problem and dividing by the number of questions. A high score indicates that symptoms are severe and functional capacity is limited. The maximum score on this scale is 40 and the minimum score is 8.
The electrophysiological examination | end of 1. month
  The electrophysiological examination was performed using the Nihon Koden Neuropack 2- MEB 7102-K device. During the electrophysiological studies, the room temperature was set at 25 C° and the temperature of the extremities was set above 32 C˚. In our study, the standard data obtained by Oh et al. were used [17]. In the study of motor conduction of the median nerve, a superficial rod electrode was used for recording at the abductor pollicis brevis muscle. The wrist and antecubital fossa were stimulated 6 cm proximal to the recording electrode. The combined muscle action potential (CMAP) (mV) and distal motor latency (msec) were recorded. Sensory conduction was examined by orthodromic stimulation at the 2nd finger and recording at the wrist with a superficial rod electrode. The conduction velocity of the sensory action potential (SAP) was recorded.
The ultrasound examination | end of 1. month
  The ultrasound examination was performed with a Logiq 9 (GE Medical Systems®). During the ultrasound examination, the patient was in a sitting position, arms next to the body, the elbow in 90° flexion, the forearm in supination. The cross-sectional area of the median nerve and the minor and major axes were calculated using the available programme of the ultrasound machine. The echogenic line around the nerve was not considered, and a manual drawing was made along the nerve border around the hyperechoic epineurium. From the level of the proximal carpal tunnel (distal wrist line), the scaphoid and carpal bones were determined as landmarks, and the cross-sectional area of the median nerve and the major and minor axes were measured. The flattening ratio resulting from dividing the major axis by the minor axis was recorded.

SECONDARY OUTCOMES:
The Boston Symptom Severity Scale (BSSS) | end of 3. month
  The Boston Symptom Severity Scale consists of 11 questions, with each question scored between 1 and 5. The average score is calculated by summing the points received for each problem and dividing by the number of questions. A high score indicates that symptoms are severe and functional capacity is limited.The maximum score on this scale is 55 and the minimum score is 11.
The Boston Functional Capacity Scale (BFCS) | end of 3. month
  The Boston Functional Capacity Scale consists of 8 questions, with each question scored between 1 and 5. The average score is calculated by summing the points received for each problem and dividing by the number of questions. A high score indicates that symptoms are severe and functional capacity is limited. The maximum score on this scale is 40 and the minimum score is 8.
The electrophysiological examination | end of 3. month
  The electrophysiological examination was performed using the Nihon Koden Neuropack 2- MEB 7102-K device. During the electrophysiological studies, the room temperature was set at 25 C° and the temperature of the extremities was set above 32 C˚. In our study, the standard data obtained by Oh et al. were used [17]. In the study of motor conduction of the median nerve, a superficial rod electrode was used for recording at the abductor pollicis brevis muscle. The wrist and antecubital fossa were stimulated 6 cm proximal to the recording electrode. The combined muscle action potential (CMAP) (mV) and distal motor latency (msec) were recorded. Sensory conduction was examined by orthodromic stimulation at the 2nd finger and recording at the wrist with a superficial rod electrode. The conduction velocity of the sensory action potential (SAP) was recorded.
The ultrasound examination | end of 3. month
  The ultrasound examination was performed with a Logiq 9 (GE Medical Systems®). During the ultrasound examination, the patient was in a sitting position, arms next to the body, the elbow in 90° flexion, the forearm in supination. The cross-sectional area of the median nerve and the minor and major axes were calculated using the available programme of the ultrasound machine. The echogenic line around the nerve was not considered, and a manual drawing was made along the nerve border around the hyperechoic epineurium. From the level of the proximal carpal tunnel (distal wrist line), the scaphoid and carpal bones were determined as landmarks, and the cross-sectional area of the median nerve and the major and minor axes were measured. The flattening ratio resulting from dividing the major axis by the minor axis was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sidar Burcu Ates Demiroglu, Principal Investigator — Ankara Bilken City Hospital
Locations (1):
- Ankara City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Padua L, Coraci D, Erra C, Pazzaglia C, Paolasso I, Loreti C, Caliandro P, Hobson-Webb LD. Carpal tunnel syndrome: clinical features, diagnosis, and management. Lancet Neurol. 2016 Nov;15(12):1273-1284. doi: 10.1016/S1474-4422(16)30231-9. Epub 2016 Oct 11. PMID 27751557
- [Background] Ezzati K, Laakso EL, Salari A, Hasannejad A, Fekrazad R, Aris A. The Beneficial Effects of High-Intensity Laser Therapy and Co-Interventions on Musculoskeletal Pain Management: A Systematic Review. J Lasers Med Sci. 2020 Winter;11(1):81-90. doi: 10.15171/jlms.2020.14. Epub 2020 Jan 18. PMID 32099632
- [Background] Cheung WKW, Wu IXY, Sit RWS, Ho RST, Wong CHL, Wong SYS, Chung VCH. Low-level laser therapy for carpal tunnel syndrome: systematic review and network meta-analysis. Physiotherapy. 2020 Mar;106:24-35. doi: 10.1016/j.physio.2019.06.005. Epub 2019 Jun 20. PMID 32026843
- [Background] Hojjati F, Afjei MH, Ebrahimi Takamjani I, Rayegani SM, Sarrafzadeh J, Raeissadat SA, Payami S. The Effect of High-Power and Low-Power Lasers on Symptoms and the Nerve Conduction Study in Patients With Carpal Tunnel Syndrome. A Prospective Randomized Single-Blind Clinical Trial. J Lasers Med Sci. 2020 Fall;11(Suppl 1):S73-S79. doi: 10.34172/jlms.2020.S12. Epub 2020 Dec 30. PMID 33995973